CLINICAL TRIAL: NCT04627649
Title: Accuracy of Complete-arch Digital Implant Impression With Newly Designed Scan Bodies
Brief Title: Accuracy of Digital Implant Impression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhuofan Chen, Professor, Sun Yat-sen University
Other Study IDs: RuoxuanHuang
Record Dates: First submitted 2020-10-19; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Edentulous Jaw
Keywords: dental implant; digital impression; scan body; accuracy
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the accuracy of complete-arch digital implant impression using newly designed scan bodies with extensional structure.

DETAILED DESCRIPTION:
Fully edentulous patients with 2-6 dental implants are included in this study. For each patient, the follow three impressions are made: conventional splinted open-tray impression, digital impression using scan bodies without extensional structure, and digital impression using scan bodies with extensional structure. The accuracy of the three impressions is compared in an inspection software.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and able to understand an informed consent
* Fully edentulous jaw
* 2-6 dental implants have been placed in the edentulous jaw
* The implants have been osseointegrated
* Mouth opening larger than 4.5 cm

Exclusion Criteria:

* Poor oral hygiene
* Presence of peri-implantitis or peri-implant mucositis
* Presence of temporamandibular joint disease
* Unwilling to paticipate in the research

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 patients are anticipated.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
accuracy | 0 day
  the accuracy is evaluated by comparing the test scans with the reference scan

CONTACTS AND LOCATIONS:
Overall Officials: Zhuofan Chen, DDS, Study Director — Guanghua School of Stomatology, Hospital of Stomatology, Sun Yat-sen University
Locations (1):
- Guanghua school of stomatology, hospital of stomtology, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chochlidakis K, Papaspyridakos P, Tsigarida A, Romeo D, Chen YW, Natto Z, Ercoli C. Digital Versus Conventional Full-Arch Implant Impressions: A Prospective Study on 16 Edentulous Maxillae. J Prosthodont. 2020 Apr;29(4):281-286. doi: 10.1111/jopr.13162. Epub 2020 Mar 24. PMID 32166793
- [Background] Mizumoto RM, Yilmaz B, McGlumphy EA Jr, Seidt J, Johnston WM. Accuracy of different digital scanning techniques and scan bodies for complete-arch implant-supported prostheses. J Prosthet Dent. 2020 Jan;123(1):96-104. doi: 10.1016/j.prosdent.2019.01.003. Epub 2019 Apr 27. PMID 31040026

DOCUMENTS (1):
  • Study Protocol (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04627649/Prot_000.pdf